CLINICAL TRIAL: NCT06835504
Title: Efficacy of Intravenous Sub-Dissociative Ketamine Versus Intravenous Morphine in Children With Acute Pain
Brief Title: Morphine or Ketamine for Analgesia
Acronym: MoKA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Daniel S Tsze, MD, MPH, Professor of Pediatrics in Emergency Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAV7115; U01HD116253 (NIH); IRB00181652 (Other: University of Utah Institutional Review Board)
Record Dates: First submitted 2024-12-16; First posted 2025-02-19 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Abdominal Pain; Isolated Extremity Fracture; Pain; Pediatrics
Keywords: Ketamine; Morphine; Pediatric; Children; Sub-dissociative; Opioid-sparing; Emergency medicine; Emergency care; Emergency department; Post-traumatic stress; Anxiety; Depression; Abdominal pain; Fracture; Analgesia
MeSH Terms: conditions — Abdominal Pain; Pain; Emergencies; Anxiety Disorders; Depression; Fractures, Bone; Agnosia | interventions — Ketamine; Morphine

STUDY DESIGN:
Intervention Model Description: Non-inferiority trial design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sub-dissociative ketamine (Experimental): 0.25 mg/kg, maximum dose 25 mg
  Interventions: Drug: Ketamine hydrochloride
- Morphine (Active Comparator): 0.1 mg/kg, maximum dose 8 mg
  Interventions: Drug: Morphine sulphate

INTERVENTIONS:
Drug: Ketamine hydrochloride — Sub-dissociative ketamine, IV
  Arms: Sub-dissociative ketamine
Drug: Morphine sulphate — Morphine, IV
  Arms: Morphine

SUMMARY:
Pain is common in children presenting to the emergency department but is frequently undertreated, leading to both short- and long-term consequences. Morphine is the standard treatment for children with moderate to severe acute pain, but its use is associated with serious side effects and caregiver and clinician concerns related to opioid administration. The investigators aim to determine if sub-dissociative ketamine is non-inferior to morphine for treating acute pain and a preferable alternative for treating acute pain in children because of its more favorable side effect profile and potential long-term benefits related to pain-related function, analgesic use/misuse, and mental and behavioral health outcomes.

DETAILED DESCRIPTION:
Aim 1: To determine if IV sub-dissociative ketamine is non-inferior to IV morphine for decreasing pain intensity in children presenting to an ED with acute pain. The investigators hypothesize that IV sub-dissociative ketamine is non-inferior to IV morphine for decreasing pain intensity in children with acute abdominal pain or an extremity fracture.

Aim 2: To compare the rate of acute (<2 hours) adverse events, including cardiopulmonary adverse events, associated with IV sub-dissociative ketamine and IV morphine. The investigators hypothesize that there is a smaller proportion of cardiopulmonary adverse events associated with IV sub-dissociative ketamine compared to IV morphine.

Aim 3: To determine the relationship between ketamine and long-term sequelae of acute pain. The investigators hypothesize that children who receive ketamine will have better levels of pain-related function during the first week following ED presentation and will have greater odds of experiencing more favorable post-traumatic stress, anxiety and depression outcomes 1-6 months after ED presentation compared to children who received IV morphine.

ELIGIBILITY:
Inclusion Criteria:

1. Abdominal pain or isolated long-bone extremity fracture (suspected or proven)
2. Self-reported pain score of ≥ 6/10
3. Requires IV morphine for analgesia as determined by the treating physician

Exclusion Criteria:

1. Weight > 82.4 kg
2. Known allergy/contraindication to morphine or ketamine
3. Antecedent receipt of ketamine related to presenting complaint
4. Inability to use self-report measures of pain or questionnaires
5. Chronic disease associated with pain
6. Chronic pain condition requiring use of opioids as outpatient
7. Hemodynamic instability or critical illness per treating physician
8. Altered mental state (e.g., GCS , 14 or clinical intoxication)
9. Known history of schizophrenia, liver or kidney problems, or osteogenesis imperfecta
10. Concern for open fracture, neurovascular compromise, or compartment syndrome
11. Injuries in addition to the extremity injury (e.g., head, neck, abdomen)
12. Known or reported pregnancy
13. Does not speak English or Spanish
14. Patient previously enrolled in this study
15. Wards of state, foster children, or children in custody

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1010 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Up to 120 minutes after completion of study drug administration or until a terminal event occurs
  Self-reported pain intensity measured using the Verbal Numerical Rating Scale (VNRS). Scored from 0 to 10. A higher score indicates a worse outcome.
Adverse events, acute | Up to 120 minutes after completion of study drug administration or until a terminal event occurs
  Examples of adverse events include, but are not limited to, cardiopulmonary adverse events (e.g., hypoxia, respiratory depression, hypotension); opioid-related adverse events; and adverse events as measured using the Side Effects Rating Scale of Dissociative Anesthetics (SERSDA).
Pain-related function | Days 1, 2,3, 7 and 30 after discharge.
  Pain intensity and related functional limitations due to pain, measured using the Parents' Postoperative Pain Measure (PPPM). Scored from 0 to 10. A higher score indicates a worse outcome.
Traumatic stress, primary assessment | Baseline (at time of enrollment) and days 7, 30, 90 and 180 after discharge.
  Stress related to the pain experienced measured using the Child Stress Disorder Checklist (CSDC-SF). Scored from 0 to 8. A higher score indicates a worse outcome.

SECONDARY OUTCOMES:
Receipt of rescue analgesia | Up to 120 minutes after completion of study drug administration or until a terminal event occurs
  Number of participants who received a rescue analgesic administered.
Desire for same analgesic | At 240 minutes after completion of study drug administration or when a terminal event occurs
  Number of participants who would want the same analgesic (i.e., study medication) again in the future.
Depth of sedation | Up to 120 minutes after completion of study drug administration or until a terminal event occurs
  Depth of sedation measured using the University of Michigan Sedation Scale (UMSS). Scored from 0 to 4. 0 is deepest level of sedation (unarousable), 4 is awake and alert.
Analgesic/opioid use after discharge | Days 1, 2, 3, 7, 30, 90, and 180 after discharge
  Name, dose and duration of analgesics and/or opioids used to calculate total days of use during the elapsed time since last assessment
Missed school or work | Day 7, 30, 90, 180 after discharge
  Days of missed school or work related to the chief complaint.
Return visit | Day 7, 30, 90, 180 after discharge
  Number of return visits related to the chief complaint, which can include (but not limited to) return visits to the emergency department or primary care physician
Anxiety | Baseline (at time of enrollment) and days 7, 30, 90, and 180 after discharge
  General Anxiety Disorder-7 (GAD-7). Scored from 0 to 21. A higher score indicates a worse outcome.
Depression | Baseline (at time of enrollment) and days 7, 30, 90, and 180 after discharge
  Patient-Reported Outcomes Measurement Information System (PROMIS). Scored from 8 to 40. A higher score indicates a worse outcome.
Substance use | Baseline (at time of enrollment) and days 7, 30, 90, and 180 after discharge
  National Institute on Drug Abuse (NIDA) modified assist tool. Scored from 0 to 360. A higher score indicates a worse outcome.

OTHER OUTCOMES:
Global satisfaction | Up to 120 minutes after completion of study drug administration or until a terminal event occurs
  Global satisfaction with analgesia measured using the Patient Global Impression of Change (PGIC) score. Scored from 1 to 7. A higher score indicates a worse outcome.
Opioid use/misuse | Days 30, 90, and 180 after discharge
  Name, dose and duration of opioids used to calculate total days of use during the elapsed time since last assessment and indication for use
Pain catastrophizing | Baseline (at time of enrollment) and day 7 after discharge.
  Assessment of heightened negative cognitive and affective pain responses in children. Measured using the Pain Catastrophizing Scale (PCS) for Children. Scored from 0 to 4. A higher score indicates more catastrophizing.
Pain interference | Day 7 after discharge
  How much pain interferes with daily activities measured using the Brief Pain Inventory (BPI) Pain Interference. Scored from 0 to 10. A higher score indicates a worse outcome.
Physical functioning | Baseline (at time of enrollment) and day 7 after discharge
  Health related quality of life measured using the Pediatric Quality of Life (PedsQL) inventory. Scored from 0 to 100. A higher score indicates a better health-related quality of life.
Sleep | Baseline (at time of enrollment) and day 7 after discharge
  Impact of pain on sleep measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Sleep Disturbance 8a + sleep duration. Scored from 8 to 40. A higher score indicates a worse outcome.
Traumatic stress, secondary assessment | Days 7, 30, 90, and 180 after discharge.
  University of California Los Angeles Post-Traumatic Stress Disorder (UCLA PTSD). Scored from 0 to 108. A higher score indicates a worse outcome.
Parent/Guardian/Caregiver Pain Catastrophizing | Day 180 after discharge
  Pain Catastrophizing Scale (PCS) for Parents. Scored from 0 to 52. A higher score indicates a worse outcome.
Parent/Guardian/Caregiver Pain Depression | Day 180 after discharge.
  Patient Health Questionnaire-2 (PHQ-2). Scored from 0 to 6. If the score is 3 or greater, major depressive disorder is likely.
Parent/Guardian/Caregiver Pain Anxiety | Day 180 after discharge
  Generalized Anxiety Disorder 2-item (GAD-2). Scored from 0 to 6. A higher score indicates a worse outcome.
Parent/Guardian/Caregiver Pain Quality of Life | Day 180 after discharge
  World Health Organization Quality of Life-2 item (WHOQOL-2). Scored from 2 to 10. A higher score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Tsze, MD, MPH, Principal Investigator — Columbia University; Amy L Drendel, DO, MS, Principal Investigator — Medical College of Wisconsin
Locations (8):
- United States (8):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UC Davis Children's Hospital, Sacramento, California
  - Nemours Children's Hospital, Wilmington, Delaware
  - Arthur M. Blank Hospital, Atlanta, Georgia
  - NewYork Presbyterian Morgan Stanley Children's Hospital, New York, New York
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Consistent with the HEAL Public Access and Data Sharing Policy, one of our goals is to assure rapid data sharing. The de-identified Underlying Primary Data will only be shared when confirmed to be de-identified by the EMSC Data Center (EDC), according to the standards set forth in the Department of Health and Human Services Regulations for the Protection of Human Subjects, to ensure that the identities of research participants cannot be readily ascertained from the data. Underlying Primary Data will also be stripped of identifiers according to the HIPAA Privacy Rule. The EDC is familiar with these processes given their vast experience with data management. The de-identified data will be made available at the conclusion of the project period, and any manuscripts published before the end of the project period will have accompanying release of relevant deidentified data at the time of the manuscript publications.
Supporting Information: Study Protocol, SAP
Time Frame: The de-identified data will be made available at the conclusion of the project period (currently August 2029, but may be subject to an extension), and any manuscripts published before the end of the project period will have accompanying release of relevant deidentified data at the time of the manuscript publications. The investigators recognize that the NIH may require a particular repository to be used, but otherwise, the investigators intend to submit the end-of-study data to NICHD DASH, in which case the end date of access would be subject to NICHD DASH policies.
Access Criteria: Because it is a condition of the NIH for newly funded studies to make data publicly available, the investigators are not sure what the future use may be. For our intended repository (NICHD DASH), applicants to receive the releasable data are required to abide by the User Agreement. The investigators note that if there are published manuscripts before the project period ends, minimal de-identified data would be made available to support the manuscript's reproducibility and enable further work. Such pre-trial-completion releases of deidentified data are to comply with Helping to End Addiction Long-term (HEAL) policies on data availability. The end-of-study deidentified data will be findable and available through the NICHD DASH repository's search functionality. The investigators will also note where the data are available in the primary study manuscript; as required for HEAL Initiative®-funded trials, the publications from this trial will be available as open access.
URL: https://dash.nichd.nih.gov/resource/DASHUserAgreement